CLINICAL TRIAL: NCT01944254
Title: Comparison of the Precision of Cardiac Output-measures at Random to Respiration, Synchronised With Expiration and Instructed Slow Exhalation, Obtained by Pulmonal Artery Catheter Thermodilution Technique With Cold Injection
Brief Title: The Precision of Pulmonary Artery Cardiac Output-measurements in Spontaneously Breathing Patients
Acronym: TEMP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013/409
Record Dates: First submitted 2013-09-07; First posted 2013-09-17 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Heart Diseases
Keywords: Cardiac surgical procedures; Pulmonary Artery Catheterizations; Cardiac output; Swan Ganz Catheterization
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- random to respiration (Active Comparator): Cardiac output measurement at random to respiration
  Interventions: Procedure: Cardiac output measurement at random to respiration
- timed with expiration start (Experimental): Cardiac output measurement synchronised at start of expiration.
  Interventions: Procedure: Cardiac output measurement synchronised at start of expiration
- timed to instructed exhalation (Experimental): Cardiac output measurement timed to instructed exhalation. The patient will receive instructions to exhale slowly using a peak expiratory flow (PEF)-flute and the cardiac output measurement will be started (i.e bolus given) at the start of expiration.
  Interventions: Procedure: Cardiac output measurement timed to instructed exhalation

INTERVENTIONS:
Procedure: Cardiac output measurement at random to respiration — Cardiac output measurement obtained by pulmonary artery catheter thermodilution technique (PAC TD)
  Arms: random to respiration
Procedure: Cardiac output measurement synchronised at start of expiration — Cardiac output measurement obtained by PAC TD
  Arms: timed with expiration start
Procedure: Cardiac output measurement timed to instructed exhalation — Cardiac output measurement obtained by PAC TD
  Arms: timed to instructed exhalation

SUMMARY:
The intention of this study is to determine whether the precision of the measure of cardiac output can be optimized by conducting the measurement while the participant is instructed to exhale slowly. This will be compared to measurements done at random to respiration and timed with the participant's spontaneous expiration.

ELIGIBILITY:
Inclusion Criteria:

* Every patient that receives a pulmonary artery catheter (PAC) related to elective cardiac surgeries,
* informed and written consent to participation in the study in accordance with the Helsinki declaration
* hemodynamic stability

Exclusion Criteria:

* Hemodynamical instability
* atrial fibrillation
* tricuspid insufficiency ≥ grade 2
* hemodialysis or other conditions where extra volume load can be negative,
* lack of ability to give a written consent to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The observed variance amongst the cardiac output measures | 1 hour
  The measures will be obtained the first postoperative morning by pulmonary artery catheter thermodilution technique. In total 24 measurements will be done in each patient, i.e 8 measurements in each interventional series described later. The variance observed will create the foundation for calculating the precision of the measures.

CONTACTS AND LOCATIONS:
Overall Officials: Idar Kirkeby-Garstad, Dr., Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of circulation and medical imaging, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Kjetsa E, Skjaervold NK, Skogvoll E, Kirkeby-Garstad I. Synchronizing thermodilution cardiac output measurements with spontaneous breathing does not improve precision. Acta Anaesthesiol Scand. 2016 Mar;60(3):354-9. doi: 10.1111/aas.12650. Epub 2015 Oct 26. PMID 26497869